CLINICAL TRIAL: NCT03772327
Title: HIV Adherence Bottle Intervention Trial (HABIT)
Brief Title: HIV Adherence Bottle Intervention Trial
Acronym: HABIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: AdhereTech (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1308014206
Record Dates: First submitted 2018-11-26; First posted 2018-12-11 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: HIV-1-infection; Adherence, Medication
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine counseling + AdhereTech bottle (Experimental): Participants will receive routine medication adherence counseling and be given the AdhereTech "smart bottle" with reminders.
  Interventions: Device: Adheretech "smart bottle"; Behavioral: Routine adherence counseling
- Routine counseling (Active Comparator): Participants will receive routine medication adherence counseling.
  Interventions: Behavioral: Routine adherence counseling

INTERVENTIONS:
Device: Adheretech "smart bottle" — A "smart pill bottle" that measures the exact number of pills in the bottle in real-time, sends this HIPAA-compliant data to a central server, and based on the results, can remind participants to take their medication through a phone call or text message.
  Arms: Routine counseling + AdhereTech bottle
Behavioral: Routine adherence counseling — Participants will be provided with routine adherence counseling

SUMMARY:
This is a randomized study for participants treated with tenofovir-based antiretroviral drug regimens with a history of suboptimal adherence (detectable HIV RNA twice over the last year). Eligible participants are enrolled, receive routine adherence counseling and are randomized to receive an AdhereTech "smart pill bottle" or not (open label). The "smart pill bottle" quantitates the number of tenofovir-containing pills taken and sends this to a centralized server; if a dose is missed, the participant is contacted by either phone or text. Participants are assessed at baseline and weeks 4, 8, and 12 for tenofovir diphosphate (TFV-DP) levels (by plasma and dried red blood cell spots), HIV RNA level, and adherence using a standardized questionnaire. Primary outcome is change in TFV-DP levels from baseline in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Taking a tenofovir-containing antiretroviral regimen for HIV treatment
* Documented suboptimal adherence (2 HIV RNA levels documented above the level of detection, i.e. not suppressed, on 2 occasions over the prior 52 weeks

Exclusion Criteria:

* Plans to change the current HIV drug regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy M Gulick, MD, MPH, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ellsworth GB, Burke LA, Wells MT, Mishra S, Caffrey M, Liddle D, Madhava M, O'Neal C, Anderson PL, Bushman L, Ellison L, Stein J, Gulick RM. Randomized Pilot Study of an Advanced Smart-Pill Bottle as an Adherence Intervention in Patients With HIV on Antiretroviral Treatment. J Acquir Immune Defic Syndr. 2021 Jan 1;86(1):73-80. doi: 10.1097/QAI.0000000000002519. PMID 33306564

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred primarily from the clinic population receiving care for HIV at New York Presbyterian Hospital Center for Special Studies located in New York City. A total of 24 and 42 participants were recruited from the Upper East Side and Chelsea locations respectively from May 2015 to August 2018.
Pre-assignment Details: 67 were screened for the study and 4 did not enroll because: 1 elected not to participate given excellent adherence to medications, 1 was ineligible after a switch off a tenofovir containing regimen, 1 did not come to the enrollment appointment, and 1 did not provide consent.
Period: Overall Study
Arm/Group | Routine Counseling + AdhereTech Bottle | Routine Counseling
Started (Eligible participants were randomized at the end of a screening visit) | 30 | 33
Week 0 Visit | 28 (2 participants were lost to follow up after randomization prior to any study interventions.) | 33
Completed | 25 | 26
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Counseling + AdhereTech Bottle | Routine Counseling | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [48 to 56] | 49 [42 to 52] | 51 [43 to 55]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 23 | 23 | 46
  Female | 6 | 8 | 14
  Transgender | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 16
  Not Hispanic or Latino | 21 | 20 | 41
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 14 | 30
  White | 8 | 12 | 20
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 7 | 11
HIV RNA <= 20 copies/mL [Count of Participants; unit: Participants] | 16 | 15 | 31
CD4 [Median (Inter-Quartile Range); unit: cells/μL] | 380 [227 to 580] | 428 [306 to 616] | 409 [242 to 612]
Number of daily antiretroviral pills [Median (Inter-Quartile Range); unit: pills per day] — Population: 2 participants in the Routine counseling + AdhereTech bottle group were lost to follow up before the medication data could be collected at the baseline visit.
  pills per day
    number analyzed (Participants) | 28 | 33 | 61
    (all) | 2 [1 to 3] | 3 [1 to 3] | 3 [1 to 3]
Number of participants reporting days of no missed doses in prior 4 days [Count of Participants; unit: Participants] — In the four days prior to baseline visit the number of days on which participants reported missing no doses of antiretroviral medication Population: 2 participants in the Routine counseling + AdhereTech bottle group were lost to follow up before the adherence could be collected at the baseline visit.
  Participants
    number analyzed (Participants) | 28 | 33 | 61
    4 days | 18 | 19 | 37
    3 days | 6 | 2 | 8
    2 days | 4 | 6 | 10
    1 day | 0 | 3 | 3
    No days | 0 | 3 | 3
Number of participants prescribed a tenofovir containing regimen [Count of Participants; unit: Participants] — Population: 2 participants in the Routine counseling + AdhereTech bottle group were lost to follow up before the medication data could be collected at the baseline visit.
  Participants
    number analyzed (Participants) | 28 | 33 | 61
    (all) | 28 | 33 | 61
Number of participants prescribed a NRTI containing regimen [Count of Participants; unit: Participants] — Population: 2 participants in the Routine counseling + AdhereTech bottle group were lost to follow up before the medication data could be collected at the baseline visit.
  Participants
    number analyzed (Participants) | 28 | 33 | 61
    (all) | 28 | 33 | 61
Number of participants prescribed a NNRTI containing regimen [Count of Participants; unit: Participants] — Population: 2 participants in the Routine counseling + AdhereTech bottle group were lost to follow up before the medication data could be collected at the baseline visit.
  Participants
    number analyzed (Participants) | 28 | 33 | 61
    (all) | 6 | 7 | 13
Number of participants prescribed a Protease inhibitor containing regimen [Count of Participants; unit: Participants] — Population: 2 participants in the Routine counseling + AdhereTech bottle group were lost to follow up before the medication data could be collected at the baseline visit.
  Participants
    number analyzed (Participants) | 28 | 33 | 61
    (all) | 10 | 15 | 25
Number of participants prescribed an Integrase inhibitor containing regimen [Count of Participants; unit: Participants] — Population: 2 participants in the Routine counseling + AdhereTech bottle group were lost to follow up before the medication data could be collected at the baseline visit.
  Participants
    number analyzed (Participants) | 28 | 33 | 61
    (all) | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Tenofovir Diphosphate (TFV-DP) Drug Levels
Description: Using dried blood spots from red blood cells, TFV-DP levels will be assessed.
Time Frame: Baseline and Week 12
Population: Of the 5 in AdhereTech bottle group missing baseline TFV-DP levels 2 were lost to follow up prior to the visit and 3 are missing levels. 3 participants in AdhereTech group left the study before Week 12. 4 participants in the routine counseling group are missing TFV-DP levels from baseline visit and then 7 left the study prior to Week 12.
Measure: Median (Inter-Quartile Range); unit: fmol/punch
Arm/Group | Routine Counseling + AdhereTech Bottle | Routine Counseling
Number analyzed (Participants) | 30 | 33
fmol/punch
  Baseline: number analyzed (Participants) | 25 | 29
  Baseline | 1230 [923 to 2066] | 1108 [418 to 1886]
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 1887 [797 to 2794] | 1084 [504 to 1175]
Statistical Analysis 1: Comparison: Routine Counseling + AdhereTech Bottle vs Routine Counseling; The power calculation was based on a null hypothesis of no difference in mean tenofovir-diphosphate (TFV-DP) concentrations between baseline versus week 12. Expected baseline mean (SD): 900 (404) fmol/punch. 12 week mean (SD): 1332 (597) fmol/punch in the AdhereTech bottle arm vs. 900 (404) fmol/punch in control arm. Type 1 error = 0.05, power = 80%, a sample size of 32 per arm (64 total) based on a two-sided t-test with equal variance; Test type: Superiority; p = 0.070, t-test, 2 sided; A ratio of Week 12 to baseline TFV-DP levels was used rather than a raw difference as a ratio was normally distributed; Mean Difference (Net) = 0.333, 95% CI 2-sided [-0.028 to 0.694] — The mean difference is mean ratio (Week 12 TFV-DP level over the Week 0 TFV-DP level) in the Routine counseling + AdhereTech bottle arm less the mean ratio in the Routine counseling arm

2. Secondary Outcome: Number of Participants Completing the 12 Week AdhereTech Bottle Intervention Compared to the Routine Counseling Only Group.
Description: Feasibility of using the AdhereTech "Smart Pill Bottles" in individuals living with HIV as measured by the proportion of participants that complete the study compared between arms. A statistically lower proportion in the AdhereTech bottle arm compared to the routine counseling arm would suggest use of the bottle is not feasible.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Counseling + AdhereTech Bottle | Routine Counseling
Number analyzed (Participants) | 30 | 33
Participants | 25 | 26
Statistical Analysis 1: Comparison: Routine Counseling + AdhereTech Bottle vs Routine Counseling; The null hypothesis is that the proportion of randomized participants that complete a week 12 visit is not lower in the AdhereTech bottle arm; Test type: Equivalence — Equivalence defined if a two-sided 2 sample proportion test accepts the null hypothesis with p > 0.05; p = 0.89, Chi-squared, Corrected; degrees of freedom = 1; Difference in proportions = 0.045, 95% CI 2-sided [-0.179 to 0.270] — This is the proportion of those completing a week 12 visit less those completing a week 0 visit

3. Secondary Outcome: Change in Quantitative HIV Viral Load
Description: Comparative changes in quantitative HIV viral load between baseline and Week 12 in the AdhereTech bottle arm versus the routine counseling only arm.
Time Frame: Baseline and Week 12
Population: 5 and 7 participants left the AdhereTech bottle and routine counseling groups respectively. And additional participant in the AdhereTech bottle group is missing the Week 12 HIV viral load.
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | Routine Counseling + AdhereTech Bottle | Routine Counseling
Number analyzed (Participants) | 30 | 33
copies/mL
  Baseline | 19 [19 to 71] | 28 [19 to 275]
  Week 12: number analyzed (Participants) | 24 | 26
  Week 12 | 19 [19 to 49] | 26 [19 to 406]
Statistical Analysis 1: Comparison: Routine Counseling + AdhereTech Bottle vs Routine Counseling; Null hypothesis: Mean HIV viral load is not significantly different in the AdhereTech bottle group compared to the routine counseling only group; Test type: Superiority; p = 0.328, Kruskal-Wallis; Log transformation of viral load; Median Difference (Net) = -0.07 — Difference of log viral load at Week 12 less the log viral load at baseline

4. Secondary Outcome: Number of Participants With HIV RNA ≥ 20 Copies/mL at Baseline That Had a Decrease in HIV RNA to < 20 Copies/mL at Week 12 in the AdhereTech Bottle Arm Versus the Routine Counseling Only Arm.
Description: This is a measure of qualitative HIV RNA outcome. The number of participants "converting" from "detectable" (HIV RNA ≥ 20 copies/mL) at baseline to "undetectable" (HIV RNA < 20 copies/mL) at week 12 in the AdhereTech bottle arm versus the routine counseling only arm.
Time Frame: Baseline and Week 12
Population: 5 and 7 participants left the AdhereTech bottle and routine counseling groups respectively. An additional participant in the AdhereTech bottle group is missing the Week 12 HIV viral load.
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Counseling + AdhereTech Bottle | Routine Counseling
Number analyzed (Participants) | 24 | 26
Participants | 3 | 7
Statistical Analysis 1: Comparison: Routine Counseling + AdhereTech Bottle vs Routine Counseling; Null hypothesis: There is no difference in proportion of participants that go from HIV RNA ≥ 20 copies/mL to HIV RNA < 20 copies/mL between baseline to Week 12 in the AdhereTech bottle group compared the routine counseling group; Test type: Superiority; p = 0.294, Fisher Exact; Odds Ratio (OR) = 0.395, 95% CI 2-sided [0.058 to 2.044] — Odds ratio for change from HIV RNA ≥ 20 copies/mL at baseline to HIV RNA < 20 copies/mL at week 12 due to the intervention (AdhereTech bottle)

5. Secondary Outcome: TFV-DP Plasma Levels
Description: Assess TFV-DP plasma levels to compare to dried blood spot levels
Time Frame: Baseline and Week 12
Population: Funding was not obtained to obtain TFV-DP plasma levels in the study
Arm/Group | Routine Counseling + AdhereTech Bottle | Routine Counseling
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Reporting 100% Adherence to Antiretroviral Medications in During to the Prior 4 Days at Week 12.
Description: Analyze participant's self-reported adherence using National Institutes of Health AIDS Clinical Trials Group (ACTG) standardized and validated questionnaire of number of days with no missed doses of medication over prior 4 days (minimum 0, maximum 4). Number of days with missed doses was dichotomized to "no missed doses" (100% adherence) and "≥ 1 missed dose."
Time Frame: Week 12
Population: 5 and 7 participants dropped out between baseline and week 12 in the AdhereTech bottle arm and routine counseling only arms respectively. One participant in the AdhereTech bottle arm did not fully complete the adherence questionnaire at week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Counseling + AdhereTech Bottle | Routine Counseling
Number analyzed (Participants) | 24 | 26
Participants | 18 | 20
Statistical Analysis 1: Comparison: Routine Counseling + AdhereTech Bottle vs Routine Counseling; Null hypothesis: Adherence in the AdhereTech bottle arm is not better than the control arm at Week 12; Test type: Superiority; p = 1, Chi-squared, Corrected; Difference in proportions = 0.019, 95% CI 2-sided [-0.237 to 0.276]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Routine Counseling + AdhereTech Bottle | Routine Counseling
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 0/30 | 0/33

LIMITATIONS AND CAVEATS:
Unmet recruitment goals. Unexpectedly high TFV-DP dried blood spot levels in 3 participants due to unexpected drug-drug interactions. 2 participants were switched from tenofovir disproxil fumarate to tenofovir alefenamide during study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT03772327/Prot_SAP_000.pdf